CLINICAL TRIAL: NCT01228071
Title: Assessment of Time to Eugonadal Testosterone Range After Initial Fortesta (Testosterone) Gel 2% Application, Time to Steady State After Initiation of Fortesta, And Gel Drying Time After Fortesta Application
Brief Title: Time to Eugonadal Range, Time to Steady State and Drying Time
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3350-302
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Male Hypogonadism
Keywords: testosterone deficiency; hypogonadism
MeSH Terms: conditions — Eunuchism; Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 40 mg daily dose of testosterone gel 2% (Experimental): testosterone gel 2%
  Interventions: Drug: testosterone gel 2%

INTERVENTIONS:
Drug: testosterone gel 2% — 40 mg testosterone gel 2%
  Other Names: EN3350

SUMMARY:
This is a multicenter, open-label, single arm trial to evaluate the time to eugonadal testosterone range after initial testosterone gel 2% application, time to steady state after after initiation of testosterone gel 2%, and drying time after application of testosterone gel 2%.

DETAILED DESCRIPTION:
Assessment of Time to Eugonadal Testosterone Range After Initial Fortesta (Testosterone) Gel 2% Application, Time to Steady State After Initiation of Fortesta, And Gel Drying Time After Fortesta Application

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 to 65 years.
2. Have a diagnosis of primary or secondary hypogonadism with a:

   * Single morning serum total testosterone concentration <250 ng/dL or
   * Two (2) consecutive morning serum total testosterone concentrations <300 ng/dL (determined at least 1 week apart during a 3 week screening period) Total serum testosterone sampling must occur between 7 AM and 11 AM at screening
3. Have a body mass index (BMI) ≥22 kg/m2 and ≤35 kg/m2.
4. Have a hematocrit level ≤50% at screening
5. Use of reliable contraception for subjects who have sexual partners of childbearing potential (women not of childbearing potential are defined as postmenopausal, ie, amenorrhea ≥1 year or permanently sterile). Reliable methods of contraception are:

   * Barrier type devices (eg, condom, female condom, diaphragm, contraceptive sponge) only in combination with a spermicide.
   * Intra-uterine devices.
   * Oral, injectable, transdermal or implantable hormonal contraceptives.
6. Is able to understand and give written informed consent

Exclusion Criteria:

1. Severe concomitant illness, which in the opinion of the Investigator, may put the subject at risk when participating in the trial or may influence the results of the trial or affect the subjects' ability to take part in the trial.
2. Acute or chronic renal impairment [(Cr ≥ 1.5x ULN (upper limit of normal)].
3. Acute or chronic hepatic impairment will be excluded.
4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >2.5 × ULN (upper limit of normal).
5. Clinically significant, abnormal, baseline laboratory result(s), which in the opinion of the Investigator affect(s) the subject's suitability for the trial.
6. History of, or any existing, clinically significant cardiac disease (New York Heart Association [NYHA] Class III and IV).
7. Clinically significant electrocardiogram (ECG) abnormalities such as QTcB or QTcF ≥450 msec; or QTc ≥480 msec in subjects with bundle branch block.
8. Prostate specific antigen (PSA) level >4 ng/mL.
9. An abnormality on digital rectal examination deemed to be suspicious or worrisome for cancer, such as a nodule or asymmetric induration.
10. Severe symptomatic benign prostatic hyperplasia or International Prostate Symptom Score (IPSS) >19 (at screening).
11. Sleep apnea which is untreated, or subjects with sleep apnea which is treated (including c-PAP treatment) but in the opinion of the investigator has been clinically unstable during the 3 months prior to screening.
12. Current eczema, psoriasis, sunburn, or any other clinically significant skin condition at the application site.
13. Current abrasions at site of application.
14. Malignancy (or suspected malignancy) of any type except a basal cell carcinoma. Subjects with a history of malignancy must have a disease free status ≥5 years prior to starting study treatment. Subjects who have had prostate or breast cancer are not permitted to participate in the study.
15. Known to be sensitive and/or has had an adverse skin reaction to testosterone hormone replacement therapy or topical products containing alcohol.
16. Actively or potentially trying to start a family or requiring fertility treatment or with a spouse/partner who is pregnant.
17. Participated in any experimental drug or device study within 30 days prior to starting study treatment.
18. History of alcohol or substance abuse within the last year.
19. Taking opioids for any reason within 3 days of screening
20. Receiving the following medications:

    * Androgen treatments.
    * Androgen antagonists.
    * Application of any lotions, ointments, or steroids to the application site.
    * 5alpha-reductase inhibitors (eg, finasteride, dutasteride).
21. Any subjects receiving testosterone hormone replacement treatments must abide by the indicated washout period prior to screening total serum testosterone measurement

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Connecticut Clinical Research, Middlebury, Connecticut
  - Compass Research East, LLC, Oviedo, Florida
  - Southeastern Research Group, Inc., Tallahassee, Florida
  - Men's Health Boston, Brookline, Massachusetts
  - Tory Internal Medicine, PC, Troy, Michigan
  - Matrix Research, LLC, Greer, South Carolina
  - Cetero Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, open-label, single-arm phase 3B trial was initiated on November 9, 2010 and completed on May 6, 2011 in the United States.
Pre-assignment Details: After the 3-week screening period and fulfilling the eligibility criteria, 34 hypogonadal men were enrolled in the study.
Groups:
- 40 mg Daily Dose of Testosterone Gel 2%: testosterone gel 2%
  testosterone gel 2% : 40 mg testosterone gel 2%
Period: Overall Study
Arm/Group | 40 mg Daily Dose of Testosterone Gel 2%
Started | 34
Completed | 32
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic (PK) population consisted of all subjects who had a drug drying time, required trough concentrations values, and no protocol violations significantly affecting the PK data. All subjects who received at least 1 dose of study drug were included in the safety population.
Arm/Group | 40 mg Daily Dose of Testosterone Gel 2%
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Time to Target Eugonadal Range
Description: The time to eugonadal range (ie, testosterone ≥300 ng/dL) was assessed based on the 24-hour PK serum concentration data.
Time Frame: 24 hours
Population: Of the 31 subjects in the PK population, 7 subjects were not included in the analysis for time to eugonadal range. Five (5) subjects had total testosterone serum concentrations of ≥300 ng/dL at Visit 2 (baseline, time 0) and 2 subjects had total testosterone serum concentrations that never reached 300 ng/dL.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | 40 mg Daily Dose of Testosterone Gel 2%
Number analyzed (Participants) | 24
hours | 2.85 [1.91 to 4.25]

2. Primary Outcome: Time to Steady State (SS)
Description: Trough total testosterone levels were obtained at Day 2, Day 3, Day 4, Day 7, and Day 14 to assess time to steady state. Trough concentrations over the 14-day period were used to calculate time SS.
Time Frame: 14 days
Population: The PK population consisted of all subjects who had a drug drying time, required trough concentrations values, and no protocol violations significantly affecting the PK data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 40 mg Daily Dose of Testosterone Gel 2%
Number analyzed (Participants) | 31
days | 1.13 [0.68 to 3.40]

3. Primary Outcome: Gel Drying Time
Description: Testosterone gel 2% drying time was assessed with a stopwatch. On Day 14 at the time of application of the gel directly to the first anteromedial thigh, the subject started a stopwatch. The gel was spread as evenly as possible over an area of 1 g/100 cm2. The total coverage area on the thigh was approximately equal to two (2) 3"× 5" postcards. The subject gently rubbed the gel with his fingertip in a circular motion (avoiding contact with the scrotal region) until the gel was dry. At this time, the stopwatch was stopped and the time expended was recorded in the eCRF.
Time Frame: 1 day; drying time measured following gel application on Day 14
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 40 mg Daily Dose of Testosterone Gel 2%
Number analyzed (Participants) | 31
minutes | 2.4 [1.7 to 3.4]

ADVERSE EVENTS:
Time Frame: Approximately two weeks plus 21 days: AE data were collected from Screening (Day -21 to Day -1) through Day 14/End of Study(EOS).
Description: All AEs were recorded in the eCRF, including any new (or increased severity of) signs, symptoms, injury, or illness. AEs that occurred up to 14 days following the last dose of study medication were recorded on the CRF/eCRF. Any AE that was ongoing at completion/termination of the study was followed until resolution or up to 14 days.
Groups:
- EN3350 (Testosterone Gel 2%): testosterone gel 2%
  testosterone gel 2% : 40 mg testosterone gel 2%
Arm/Group | EN3350 (Testosterone Gel 2%)
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 6/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EN3350 (Testosterone Gel 2%) (N=34)
Application site dryness (General disorders) | 1
Application site rash (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less